CLINICAL TRIAL: NCT04933773
Title: SpO2 Measurement Depending on Different Pulse Oximeter Averaging Time Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: POAveragingTime21
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Movement Artifacts During SpO2 Measurements; Reduced Perfusion During SpO2 Measurements
Keywords: pulse oximetry; SpO2; averaging time; motion artifacts

STUDY DESIGN:
Intervention Model Description: All participants go through all study arms, in random order. Two pulse oximeters with different averaging time settings are active simultaneously during measurement on each participant and the measured signal is compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Set averaging times: 2-4 seconds and 8 seconds (Experimental): SpO2 is measured by two pulse oximeters on one participant's hand (on the index finger and middle finger). One pulse oximeter is set to an averaging time of 2-4 seconds, the second pulse oximeter is set to an averaging time of 8 seconds.
  Interventions: Other: Movement artifact - knocking; Other: Movement artifact - tremor; Other: Artifact - ambient light; Other: Artifact - low perfusion; Other: SpO2 measurement
- Set averaging times: 8 seconds and 16 seconds (Experimental): SpO2 is measured by two pulse oximeters on one participant's hand (on the index finger and middle finger). One pulse oximeter is set to an averaging time of 8 seconds, the second pulse oximeter is set to an averaging time of 16 seconds.
  Interventions: Other: Movement artifact - knocking; Other: Movement artifact - tremor; Other: Artifact - ambient light; Other: Artifact - low perfusion; Other: SpO2 measurement

INTERVENTIONS:
Other: Movement artifact - knocking — 60 seconds motion artifact simulation - knocking with sensors
Other: Movement artifact - tremor — 60 seconds motion artifact simulation - tremor with sensors
Other: Artifact - ambient light — 60 seconds artifact simulation - ambient light using sensor opening
Other: Artifact - low perfusion — 60 seconds artifact simulation - reduced perfusion using a cuff
Other: SpO2 measurement — Two SpO2 measuring devices are active simultaneously on one hand during measurement.

SUMMARY:
The aim of this study is to characterize the noise in the SpO2 signal depending on different pulse oximeter averaging time settings.

DETAILED DESCRIPTION:
Noise in the SpO2 signal is most often caused by artifacts, such as movement artifacts, reduced perfusion, additional light and others. These artifacts can be partially removed from the SpO2 signal by different pulse oximeter settings, specifically the sensitivity mode and averaging time. It is known that when a longer averaging time is set, the measured signal contains fewer artifacts, on the other hand there is an increased risk of missing short desaturation. The aim of this work is to characterize the noise in the SpO2 signal depending on the set averaging time of the pulse oximeter based on experimental data from healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers from the Czech Technical University

Exclusion Criteria:

* pregnancy
* severe cardiovascular conditions
* injury to the upper limbs or hands that could affect the peripheral perfusion
* diabetes
* hypotension or hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
SpO2 readings with different averaging times | 30 minutes
  Differences in the SpO2 signal during artifacts depending on the set averaging time.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Rafl Huttova, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No